CLINICAL TRIAL: NCT03994159
Title: Impact of an Emotional Robot on Quality of Working Life of Caregivers in a Geriatric Unit Specialized in Dementia
Brief Title: Impact of an Emotional Robot on Quality of Working Life of Caregivers in a Geriatric Unit
Acronym: PARO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier le Mans (Other)
Collaborators: Centre Hospitalier de Chateau du Loir (Unknown); Centre Hospitalier de Saint Calais (Unknown); Centre Hospitalier Local de Beaumont sur Sarthe (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CHM-2019/S18/06.
Record Dates: First submitted 2019-06-06; First posted 2019-06-21 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Burnout, Professional; Stress; Anxiety
MeSH Terms: conditions — Burnout, Professional; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Quasi experimental before-after study, with a mixed qualitative and quantitative approach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PARO emotional robot (Experimental): Quasi-experimental before after study of the impact of the PARO robot on team dynamics among caregivers in geriatric wards caring for patients with dementia.
  Pre intervention period: no PARO robot. Post-intervention period: with the PARO robot.
  Interventions: Device: Use of the "PARO" emotional robot

INTERVENTIONS:
Device: Use of the "PARO" emotional robot — PARO is an advanced interactive therapeutic robot designed to stimulate patients with Dementia, Alzheimer's, and other cognition disorders.

SUMMARY:
Since February 2016, with the objective of improving the quality of life and the autonomy of residents, the Le Mans General Hospital uses an interactive "emotional" robot within its geriatric wards.

This emotional robot, Paro, is equipped with a dozen sensors, 3 microphones and interacts with its user: it reacts to touch, voice and heat making small sounds and moves its head, fins and tail. The algorithm that governs Paro's behavior allows him to offer a behavioral answer adapted to the user's stimuli. Thus, Paro is able to communicate beneficial emotions to patients.

To this day however there is no published study exploring the effect of such a robot on team dynamics among caregivers in hospital units.

Our research aims at highlighting the benefits that a healthcare team perceives when working with this tool among patients suffering from dementia.

ELIGIBILITY:
Inclusion Criteria:

* Non medical caregiver (nurse, nursing aid, orderly, psychological aid worker) working in one of the selected geriatric wards.

Exclusion Criteria:

* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Impact of the PARO robot on the quality of worklife among caregivers in a specialised unit dor dementia patients | 1 month
  Semidirective interviews of the caregivers about their feelings at work, before the introduction of Paro and after 1 month of use. We will use textual analysis software to reveal speech classes to avoid analysis bias and interpretation.

SECONDARY OUTCOMES:
Impact of PARO on the caregivers perception of their own health. | 1 month
  Use of the Nottingham Health Profile (NHP). The NHP consists of two parts. The first part focuses on health and comprises 38 items which deal with pain, energy, sleep, mobility, emotional reaction and social isolation. The second part focuses on life areas affected and consists of 7 items which deal with problems regarding occupation, housework, social life, family life, sexual function, hobbies and holidays. All questions have only yes/no answer options and each section score is weighted. The higher the score, the greater the number and severity of problems. The highest score in any section is 100.
Impact of PARO on the caregivers perception of their own stress at work. | 1 month
  Measure of the level of stress using the Perceived Stress Scale: 10 item questionnaire, with responses ranging from 0 to 4 for each item, with a range from 0 to 40, 0 being no perceived stress ans 40 the maximum perceived stress.
Impact of PARO on the caregivers perception of their own anxiety at work. | 1 month
  Measure of the perceived anxiety through the Hospital Anxiety and Depression Scale (HADS, a 14 item questionnaire, each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression, 0 being no perceived anxiety and 21 the maximum perceived anxiety).

CONTACTS AND LOCATIONS:
Overall Officials: Cathy LOIRAT, Principal Investigator — Centre Hospitalier du Mans
Locations (1):
- Centre Hospitalier Local Beaumont sur Sarthe, Beaumont-sur-Sarthe, France

IPD SHARING:
Plan to Share IPD: No